CLINICAL TRIAL: NCT05271214
Title: Conservative Management of Left Ventricular Assist Device Candidates
Status: Recruiting | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0574-16-TLV
Record Dates: First submitted 2022-02-26; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Advanced Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Left ventricular assist device (LVAD) candidates will be comprehensively evaluated at our center, including clinical evaluation, echocardiography, right heart catheterization, cardiopulmonary exercise test and laboratory exams. following this evaluation, patients will be treated with inotropes, diuretics, uptitrated neurohormonal therapy. vitamin and iron deficiencies will be corrected and the patients will be referred for coronary interventions and cardiac resynchronization therapy appropriately. The need for LVAD implantation will be reevaluated according to the patient's clinical condition, echocardiography and laboratory findings.

DETAILED DESCRIPTION:
Consecutive patients with advanced heart failure (HF) who will be referred for LVAD implantation starting 01/2018. All patients will have severe left ventricular systolic dysfunction (left ventricular ejection fraction < 30%) and severe HF symptoms (New York Heart Association Class III-IV), with acute or gradual decompensation of HF.

All patients will be considered candidates for LVAD implantation. As such, they will undergo extensive cardiac evaluation. This will include comprehensive echocardiography, right heart catheterization and a cardio-pulmonary exercise test. Based on this initial evaluation, patients will be graded according to the Interagency Registry for Mechanically Assisted Circulatory Support (INTERMACS) profile. Individualized guideline-directed medical therapy will be initiated. Following therapy optimization, evaluation will be repeatedly performed during the next months in order to continuously reevaluate the need for a LVAD implantation. Repeated evaluation will include clinical assessment, laboratory testing, comprehensive echocardiography and cardio-pulmonary exercise test in all cases. Repeated right heart catheterization will be done on an individual basis.

Our therapeutic goal will consist of initial stabilization during the index admission. Our protocol includes intravenous furosemide (as needed) and continuous intravenous milrinone 0.25-0.5mcg/kg/min. Intravenous thiamine (500-1,000 mg) will be added. Beta blockers will be continued or added within the first 24 hours and switched to HF-established beta blockers within 48 hours. Hydralazine will be initiated within the first 48 hours and nitrates will be added after reaching 60 mg hydralazine per day. A loading dose of digoxin (i.e. total 1mg) was given during the first 48 hours. Low dose oral digoxin with an aim of maintaining digoxin serum-levels of 0.4-0.8 ng/ml. Investigation for iron deficiency and vitamin D levels will be done within 24 hours from admission and corrections will be initiated early. Low dose spironolactone will be the first renin-angiotensin-aldosterone system inhibitor used, followed by low dose valsartan with an aim to introduce sacubitril/valsartan shortly thereafter. Type-2 sodium-glucose transporter inhibitors (SGLT2i) during the index admission will be used with an aim of decreasing diuretic doses and reach early stabilization. Coronary angiography will be routinely done and revascularization interventions will be considered on an individual basis. Cardiac resynchronization therapy (CRT) will be used when appropriate. After discharge, close follow up, at intervals of 3-14 days, will be performed at our Outpatient HF Clinic, including clinical evaluation, laboratory testing and repeated cardiac imaging. Patients will be planned to receive intravenous diuretics and inotropes (levosimendan or milrinone). Drug up-titration will be rigorously pursued.

Cardiopulmonary exercise test: Symptom-limited graded ramp exercise tests performed with the use of either bicycle ergometer (Ergoline, 100P) or treadmill ergometer (Ram, 770CE). The work-rate increment protocol is tailored to the individual to yield fatigue-limited exercise duration of about 8 to 12 min. The protocol includes 2 min of unloaded phase, a symptom-limited ramp graded exercise, and 2 min of recovery. Breath-by-breath minute tidal volume (TV), respiratory rate, VE, VCO2, and VO2 are measured using a Medical Graphics Metabolic Cart (Cortex, Metalyzer 3B). Peak VO2 is the highest averaged 30-s VO2 during exercise. Anaerobic threshold is determined manually using the modified V-slope method. VE/VCO2 slope is calculated by linear regression with all exercise data obtained from the progressive exercise test. The metabolic-chronotropic relationship is calculated from the ratio of the HR reserve to the metabolic reserve during submaximal exercise. A metabolic-chronotropic relationship slope <0.80 is considered indicative of chronotropic incompetency. In patients receiving beta-blocker therapy, chronotropic incompetency is considered to be present when <62% of HR reserve is reached.

Echocardiography: Echocardiographic evaluation performed in a standard manner, always using the same equipment (iE33, Philips Medical Systems, Bothell, WA). LVEF is calculated by Simpson's method. LV diameters, inter-ventricular septal diameter and LV posterior wall width measured during systole and diastole as recommended (8). Forward stroke volume is calculated from LV outflow tract with subsequent calculation of cardiac output. Left atrium volume is calculated using the biplane area length method at end systole. All volumetric measurements are adjusted to body surface area and reported as ml/m2. Pulsed-wave Doppler is performed in the apical 4-chamber view to obtain mitral inflow velocities to assess left ventricular filling. Recordings are averaged over 3 and ≥7 consecutive cardiac cycles during sinus rhythm and atrial fibrillation respectively. Measurements of mitral inflow included the peak early filling (E wave) and late diastolic filling (A wave) velocities, the E/A ratio, and deceleration time (DT) of early filling velocity. Early diastolic mitral annular velocities (e') measured in the apical 4-chamber view. The e' is measured from septal and lateral annulus in all studies. The ratio of peak E to peak e' (septal, lateral and average) is calculated (mitral E/e' ratio) from the average of at least 3 cardiac cycles (9). Apart from qualitative grading, right ventricular function is evaluated using S' and tricuspid annular plane systolic excursion (TAPSE). Hemodynamic assessment estimated tricuspid regurgitation velocity and right atrial pressure using the inferior vena cava to calculate the systolic pulmonary artery pressure.

Right heart catheterization. The catheterization is performed through a 7F sheath via the right internal jugular or right femoral vein. Pressures in the right atrium, right ventricle, pulmonary artery, and pulmonary capillary wedge position are measured at end expiration (mean of ≥3 beats) using fluid-filled manometer. Mean pressures are calibrated at the beginning of each case to avoid baseline drift. Transducers are zeroed at midaxillary level in each patient. Pressure tracings from the entire study are stored for offline analysis. Mean right atrium and pulmonary capillary wedged pressure (PCWP) taken at mid-A wave. PCWP position verified by typical waveforms, appearance on fluoroscopy, and, when needed, by direct oximetry (PCWP blood saturation ≥94%). Arterial blood pressure is measured noninvasively. Arterial-venous O2 content difference (AVo2diff) measured directly as the difference between systemic arterial and Pao2 content (=saturation × hemoglobin ×1.34). Oxygen consumption (Vo2) measured from expired gas analysis to calculate cardiac output (CO), by the direct Fick method (CO= Vo2÷AVo2diff).

ELIGIBILITY:
Inclusion Criteria:

- left ventricular ejection fraction <35%. New York Heart Association Class III or IV. Brain natriuretic peptide levels > 450pg/ml. Heart failure hospitalization in the past 6 months. Maximal oxygen consumption < 12 ml/kg/min. Intolerant to conventional heart failure therapy.

Exclusion Criteria:

- Special populations - pregnant, unable to give informed consent. Advanced liver disease (Child Pugh class B or C). Advanced kidney disease (eGFR<30ml/min). Severe pulmonary disease. Severe peripheral vascular disease. Active malignancy.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Advanced symptomatic heart failure patients with reduced ejection fraction in whom a left ventricular assist device implantation is planned.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
New York Heart Association (NYHA) Class | 3 months
  improvement in NYHA class

SECONDARY OUTCOMES:
Maximal oxygen consumption (VO2) | 6 months
  improvement in VO2
natriuretic peptide levels | 3 months
  reduction in brain natriuretic peptide levels
left ventricular size | 6 months
  reduction in left ventricular end diastolic diameter

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available from Dr Ofer Havakuk (oferh@tlvmc.gov.il) upon reasonable request.